CLINICAL TRIAL: NCT02836704
Title: Comparison of Efficacy and Safety of Standard vs Higher Starting Dose of Insulin Glargine in Overweight and Obese Chinese Patients With Type 2 Diabetes
Brief Title: Comparison of Standard vs Higher Starting Dose of Insulin Glargine in Chinese Patients With Type 2 Diabetes (Glargine Starting Dose)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LANTUL07191; U1111-1172-2903 (Other: UTN)
Record Dates: First submitted 2016-07-07; First posted 2016-07-19 (Estimated); Last update posted 2022-04-25 (Actual); Status verified 2022-04

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Insulin Glargine; Metformin; Acarbose

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard initial dose of insulin glargine (Active Comparator): Dose 1 of insulin glargine will be administered subcutaneously once a day at the same time every day. Previous non-sulfonylurea OADs (eg, metformin, acarbose) are background treatment and will be continued at the same dosage and dosing frequency as before.
  Interventions: Drug: INSULIN GLARGINE; Drug: metformin; Drug: acarbose
- Higher initial dose of insulin glargine (Experimental): Dose 2 of insulin glargine will be administered subcutaneously once a day at the same time every day. Previous non-sulfonylurea OADs (eg, metformin, acarbose) are background treatment and will be continued at the same dosage and dosing frequency as before.
  Interventions: Drug: INSULIN GLARGINE; Drug: metformin; Drug: acarbose

INTERVENTIONS:
Drug: INSULIN GLARGINE — Pharmaceutical form: solution
  Route of administration: subcutaneous injection
  Other Names: HOE901
Drug: metformin — Pharmaceutical form: table or capsule
  Route of administration: oral administration
Drug: acarbose — Pharmaceutical form: table or capsule
  Route of administration: oral administration

SUMMARY:
Primary Objective:

-To test the hypothesis that higher initial dose of basal insulin (0.3 U/kg) is non inferior to standard initial dose (0.2 U/kg) based on the percentage of patients with at least one episode of hypoglycemia (≤3.9 mmol/L or severe) during the 16 weeks of treatment in overweight and obese type 2 diabetic patients uncontrolled with oral anti-diabetes drugs (OADs).

Secondary Objective:

* To evaluate the percentage of patients achieving glycated hemoglobin (HbA1c) <7%.
* To evaluate the percentage and accumulated percentage of patients achieving fasting plasma glucose (FPG) target (<5.6, <6.1, and <7.0 mmol/L).
* To assess the changes in HbA1c, FPG, and postprandial glucose (PPG).
* To evaluate the insulin doses change.
* To evaluate the weight change.
* To evaluate overall hypoglycemia, nocturnal hypoglycemia and severe hypoglycemia occurrence.
* To descriptively evaluate the safety profile.
* To assess patient and physician satisfaction and adherence (drop-out rate and the percentage of patients who can follow the treatment and insulin titration).
* Subgroup analysis on efficacy (control rate, control rate without confirmed hypoglycemia, and changes in HbA1c, FPG and PPG) and safety data according to:
* Age
* Duration of diabetes
* Baseline treatment (OAD)
* Baseline HbA1c, FPG and PP

DETAILED DESCRIPTION:
The duration of study for each patient is approximately 20 weeks from screening visit to end-of-study follow-up phone call.

ELIGIBILITY:
Inclusion criteria :

* Age ≥ 18 and ≤ 70 years.
* Type 2 diabetes patients with diabetes diagnosis at least 2 years.
* Continuous treatment with stable doses of 2-3 OADs, for more than three months prior to randomization, among which metformin ≥1.5 g/day or at maximum tolerated dose
* HbA1c >7.5% and ≤11%.
* FPG >9 mmol/L.
* BMI ≥25 and ≤40 kg/m^2.
* Ability and willingness to perform self-monitoring of blood glucose using the Sponsor-provided glucose meter and to complete the patient diary.
* Willingness and ability to comply with the study protocol.
* Signed informed consent obtained prior any study procedure.

Exclusion criteria:

* Known hypersensitivity/intolerance to insulin glargine or any of its excipients.
* History of hypoglycemia unawareness.
* Unexplained hypoglycemia in the past 6 months.
* Pregnancy or planned pregnancy or current lactation (women of childbearing potential must have a negative pregnancy test at study entry and a medically approved contraception method).
* Acute diabetic complications (diabetic ketoacidosis, lactic acidosis, hyperosmolar nonketotic diabetic coma).
* History of stroke, myocardial infarction, angina pectoris, coronary artery bypass graft, or percutaneous transluminal coronary angioplasty within the previous 12 months.
* Active proliferative retinopathy, as defined by a photocoagulation or vitrectomy occurrence in the 6 months prior to study entry, or any other unstable (rapidly progressing) retinopathy that may require photocoagulation or surgical treatment during the study, documented by retina examination or disease history record, in the 2 years prior to study entry.
* Impaired renal function defined as, but not limited to, serum creatinine levels ≥1.5 mg/dL (132 μmol/L) for males and ≥1.4 mg/dL (123 μmol/L) for females or presence of macroproteinuria (>2 g/day).
* Active liver disease (alanine transaminase [ALT] greater than two times the upper limit of the reference range, as defined by the local laboratory).

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 892 (Actual)
Dates: Start 2016-09-09 (Actual); Primary Completion 2018-04-26 (Actual); Study Completion 2018-04-26 (Actual)

PRIMARY OUTCOMES:
Percentage of patients with at least one episode of hypoglycemia | 16 weeks

SECONDARY OUTCOMES:
Percentage of patients achieving HbA1c <7% | 16 weeks
Percentage of patients achieving Fasting Plasma Glucose target (<5.6, <6.1, and <7.0 mmol/L) | 16 weeks
Accumulated percentage of patients achieving Fasting Plasma Glucose target (<5.6, <6.1, and <7.0 mmol/L) | 16 weeks
Change from baseline in HbA1c | Baseline, 16 weeks
Change from baseline in Fasting Plasma Glucose | Baseline, 16 weeks
Change from baseline in Post Prandial Glucose | Baseline, 16 weeks
Change in body weight | Baseline, 16 weeks
- Change in insulin dose | Baseline, 16 weeks
Number of overall hypoglycemic events (with severe or confirmed hypoglycemia [≤3.9 mmol/L]) | Baseline, 16 weeks
Number of nocturnal hypoglycemic events | Baseline, 16 weeks
Number of severe hypoglycemic events | Baseline, 16 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (1):
- China, China

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- [Derived] Wan H, Wen B, Wang X, Wang J, Zhang Y, Ning T, Duan B, Li Y, Feng W, Zhang X, Cui N, Ji L. Effect of Baseline Characteristics on Hypoglycaemia Risk with Insulin Glargine 100 U/mL: Post Hoc Analysis of the BEYOND 7 Study. Diabetes Ther. 2021 Sep;12(9):2359-2369. doi: 10.1007/s13300-021-01112-z. Epub 2021 Jul 21. PMID 34286454
- [Derived] Ji L, Gao Z, Shi B, Bian R, Yin F, Pang W, Gao H, Cui N. Safety and Efficacy of High Versus Standard Starting Doses of Insulin Glargine in Overweight and Obese Chinese Individuals with Type 2 Diabetes Mellitus Inadequately Controlled on Oral Antidiabetic Medications (Beyond VII): Study Protocol for a Randomized Controlled Trial. Adv Ther. 2018 Jun;35(6):864-874. doi: 10.1007/s12325-018-0717-x. Epub 2018 Jun 5. PMID 29873004